CLINICAL TRIAL: NCT01086917
Title: Experimental Human Malaria Infection by Intradermal Injection of Plasmodium Falciparum Sporozoites (PfSPZ Challenge)
Brief Title: Experimental Human Malaria Infection by PfSPZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TIP2
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Malaria
Keywords: Malaria Challenge; Plasmodium falciparum; Controlled human malaria infection; PfSPZ Challenge
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): to receive a dose of 2,500 PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge
- Group 2 (Experimental): to receive a dose of 10,000 PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge
- Group 3 (Experimental): to receive a dose of 25,000 PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge

INTERVENTIONS:
Biological: PfSPZ Challenge — each volunteer to receive a single dose
  Other Names: aseptic, purified, cryopreserved Plasmodium falciparum sporozoites

SUMMARY:
The study is a single center, varied dose, open label study. A maximum of eighteen volunteers will be exposed to live NF54 P. falciparum sporozoites (PfSPZ Challenge) by intradermal injection. Volunteers will be divided into three groups of 6 volunteers, each group spaced 25 days apart (21 days after the last challenge of the last volunteer from the previous dose group).

DETAILED DESCRIPTION:
In every group on day 1, two volunteers will be injected. On day 3 the remaining four volunteers of the group will be injected. Injections in subsequent volunteers are always spaced at least one hour apart in any group. Injection of subsequent (groups of) volunteers will only commence if the previous injection was shown to be safe. Three different doses of PfSPZ will be administered: a dose of 2,500 PfSPZ Challenge (Group 1); a dose of 10,000 PfSPZ Challenge (Group 2) if not all volunteers become thick smear positive (TS+) in Group 1; and a dose of 25,000 PfSPZ Challenge (Group 3) if there is not 100% TS+ in Group 2. If all volunteers in Group 1 (2,500 PfSPZ Challenge) become thick smear positive, then Group 2a will receive 1,000 PfSPZ Challenge. If all volunteers in Group 2a become TS+, the volunteers in Group 3a will receive 500 PfSPZ Challenge. If all volunteers in Group 2 (10,000 PfSPZ Challenge) become TS+, Group 3b will receive 5,000 PfSPZ. If less than 100% of volunteers in Group 2a (1,000 PfSPZ Challenge) become TS+ then Group 3c will receive 1,750 PfSPZ Challenge.

The clinical, biological, parasitological and immunological data of these groups' volunteers will be compared. Volunteers and the investigator will not be blinded, but the laboratory personnel will be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 35 years healthy volunteers (males or females)
2. Good health based on history and clinical examination
3. Negative pregnancy test
4. Use of adequate contraception for females
5. All volunteers must sign the informed consent form demonstrating their understanding of the meaning and procedures of the study
6. Volunteer agrees to inform the general practitioner and agrees to sign a request to release medical information concerning contra-indications for participation in the study
7. Willingness to undergo a Pf sporozoite challenge
8. For volunteers not living in Nijmegen: agreement to stay in a hotel room close to the trial center during a part of the study (Day 5 till 3 days after treatment)
9. Reachable (24/7) by mobile phone during the whole study period
10. Living with a third party that could contact the clinicians in case of alteration of consciousness or agreement to stay in a hotel room close to the trial center during a part of the study (Day 5 till 3 days after treatment)
11. Available to attend all study visits
12. Agreement to refrain from blood donation to Sanquin or for other purposes, during the study period until day 140.
13. Willingness to undergo HIV, hepatitis B and hepatitis C tests
14. Negative urine toxicology screening test at screening visit and day before challenge
15. Willingness to take a curative regimen of Malarone®

Exclusion Criteria:

1. History of malaria
2. Plans to travel to malaria endemic areas during the 140 day study period
3. Plans to travel outside of the Netherlands during day 0-28 of the study
4. Previous participation in any malaria vaccine study and/or positive serology for Pf
5. Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
6. History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
7. History of arrhythmias or prolonged QT-interval
8. Positive family history in 1st and 2nd degree relatives for cardiac disease < 50 years old
9. An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
10. Clinically significant abnormalities in electrocardiogram (ECG) at screening
11. Body Mass Index (BMI) below 18 or above 30 kg/m2
12. Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
13. Positive HIV, HBV or HCV tests
14. Participation in any other clinical study within 30 days prior to the onset of the study
15. Enrollment in any other clinical study during the study period
16. Pregnant or lactating women
17. Volunteers unable to give written informed consent
18. Volunteers unable to be closely followed for social, geographic or psychological reasons
19. Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
20. A history of psychiatric disease
21. Known hypersensitivity to anti-malaria drugs
22. The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period
23. Contra-indications to Malarone® including treatment taken by the volunteer that interferes with Malarone®
24. Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia
25. Co-workers of the departments of Medical Microbiology or Internal Medicine of the Radboud University Nijmegen Medical Centre or Sanaria Inc.
26. A history of sickle cell anemia, sickle cell trait, thalassemia , thalassemia trait or G6PD deficiency

Ages: 19 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of volunteers with Plasmodium falciparum Infection | Upto 7 months
  To achieve a 100% infection rate of human volunteers by intradermal injection of aseptic, purified, cryopreserved Pf sporozoites (PfSPZ Challenge)as measured by 100% thick smear positivity (thick blood smears) of all volunteers from one group

SECONDARY OUTCOMES:
Kinetics of infection | Upto 7 months
  To compare parasite kinetics between different doses of intradermal injection of PfSPZ Challenge as measured by:
  * A significant difference in time of thick smear positivity between the groups of volunteers
  * A significant quantitative difference in parasitemia as measured by retrospective PCR between the groups of volunteers
  * A significant difference in kinetics of parasitemia between the groups of volunteers as measured by retrospective PCR
  * A difference in occurrence or intensity of signs or symptoms between the groups of volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, Md PhD, Principal Investigator — UMC St Radboud
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Roestenberg M, Bijker EM, Sim BKL, Billingsley PF, James ER, Bastiaens GJH, Teirlinck AC, Scholzen A, Teelen K, Arens T, van der Ven AJAM, Gunasekera A, Chakravarty S, Velmurugan S, Hermsen CC, Sauerwein RW, Hoffman SL. Controlled human malaria infections by intradermal injection of cryopreserved Plasmodium falciparum sporozoites. Am J Trop Med Hyg. 2013 Jan;88(1):5-13. doi: 10.4269/ajtmh.2012.12-0613. Epub 2012 Nov 13. PMID 23149582
- [Derived] Teirlinck AC, Roestenberg M, Bijker EM, Hoffman SL, Sauerwein RW, Scholzen A. Plasmodium falciparum Infection of Human Volunteers Activates Monocytes and CD16+ Dendritic Cells and Induces Upregulation of CD16 and CD1c Expression. Infect Immun. 2015 Sep;83(9):3732-9. doi: 10.1128/IAI.00473-15. Epub 2015 Jul 13. PMID 26169270